CLINICAL TRIAL: NCT01182389
Title: A Prospective Randomised Study of Early Robotic Ablation by Substrate Elimination of Ventricular Tachycardia
Brief Title: A Study of Early Robotic Ablation by Substrate Elimination of Ventricular Tachycardia
Acronym: ERASE-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Hansen Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO1631
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2016-02

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Implantable Cardioverter Defibrillator; Catheter Ablation; Robotic
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- robotic VT Ablation (Active Comparator): Robotic VT ablation by substrate elimination
  Interventions: Procedure: Robotic VT Ablation
- Conventional therapy (Active Comparator): review of ICD programming to ensure that detection and therapy will occur appropriately.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Procedure: Robotic VT Ablation — Robotic VT Ablation
  Arms: robotic VT Ablation
Other: Conventional Therapy — Review of ICD programming to ensure that detection and therapy will occur appropriately
  Arms: Conventional therapy

SUMMARY:
Ventricular tachycardia (VT) is an abnormal rapid heartbeat which occurs after a heart attack and can cause sudden death. Patients at risk of this rhythm disturbance usually receive an implantable cardioverter defibrillator (ICD) that can prevent death by returning the heart's rhythm back to normal by electrically stimulating the heart but in doing so gives the patient painful and debilitating shocks. The first ICD shock after implantation appears to be a powerful predictor of subsequent shock therapy as well as being a predictor of of increased mortality in patients with primary prevention ICDs. In patients who receive repeated shocks VT ablation is performed to 'burn' the abnormal area of the heart that causes the problem. However, it is often only performed as a last resort as it is technically challenging. We believe that performing VT ablation using the robotic system early after the first episode of VT after ICD implantation, may reduce the number of painful shocks received by the patient and possibly increase life expectancy and quality of life.

200 patients from 5 european countries will be recruited in a prospective, open, randomised trial. Eligible, consenting patients who have experienced their first episode of VT since ICD implantation, will be randomised in a 1:1 manner into treatment arms of either VT ablation or standard 'conventional' therapy and followed-up every 4 months over two years to assess the number of subsequent ICD shocks, hospitalisation, mortality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males or females eighteen (18) to eighty-five (85) years old
* ICD implantation for post-infarct primary or secondary prophylaxis
* First episode of VT detected (within monitor zone or therapy (ATP /shock delivered) or by 12 lead ECG if the rate below the detection level of the device.
* Suitable candidate for catheter ablation
* Signed informed consent

Exclusion Criteria:

* Contraindication to catheter ablation
* Ventricular tachycardia due to transient, reversible causes
* Presence of a left ventricular thrombus
* Severe cerebrovascular disease
* Active gastrointestinal bleeding
* Renal failure (on dialysis or at risk of requiring dialysis)
* Active infection or fever
* Life expectancy shorter than the duration of the trial
* Allergy to contrast
* Intractable heart failure (NYHA Class IV)
* Bleeding or clotting disorders or inability to receive heparin
* Serum [K+] <3.5 or >5.0mmol/L
* Serum Creatinine >200umol/L
* Uncontrolled diabetes (HbA1c ≥73mmol/mol or HbA1c ≤64mmol/mol and Fasting Blood Glucose ≥9.2mmol/L)
* Malignancy needing therapy
* Pregnancy or women of child-bearing potential not using a highly effective method of contraception
* Unable to give informed consent
* Unable to attend follow-up in ICD clinics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Any appropriate ICD therapy | 24 months post randomisation

SECONDARY OUTCOMES:
Treatment Failures defined as either2 ICD shocks or 5 ATP episodes | 24 months post randomisation
Total therapy rate | 24 months post randomisation
Mortality | 24 months post randomisation
All cause hospitalisation | 24 months post randomisation
Quality of Life | 12 months post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Dr Kanagaratnam, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - St Bartholomew's Hospital, London
  - Hammersmith Hospital, Imperial College Healthcare, London
  - John Radcliffe Hospital, Oxford